CLINICAL TRIAL: NCT04015440
Title: Hostile Bias Modification Training Online Study II
Acronym: HBMT II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Collaborators: Army Research Laboratory (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: WRAIR #2628
Record Dates: First submitted 2019-07-08; First posted 2019-07-11 (Actual); Results first posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Aggression; Anger; Emotion Regulation; Self-Control; Stress
Keywords: attention bias; hostile attribution bias; hostile bias modification
MeSH Terms: conditions — Aggression; Emotional Regulation; Self-Control

STUDY DESIGN:
Intervention Model Description: This is an online study. Volunteer assignment to each of the two experimental conditions is semi-randomized (i.e. random except that computer ensure equal sample sizes across experimental conditions). The randomized assigning of participants is done by the study web-page/program at volunteerscience.com. The computer program randomly assigned volunteers to one of the two conditions when they begin the study.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HBMT (Experimental)
  Interventions: Behavioral: HBMT
- Placebo (Placebo Comparator)
  Interventions: Behavioral: Other Training

INTERVENTIONS:
Behavioral: HBMT — Individual is presented with words with some letters missing and told to complete the word.
  Arms: HBMT
Behavioral: Other Training — Alternative to HBMT training
  Arms: Placebo

SUMMARY:
The purpose of this study is to see how people respond on a word completion task relates to how they behave and respond to situations in the real world. This is a two part research study. At time-point one, participants will fill out some brief personality surveys. They will also read several short scenarios and imagine how they would react and/or interpret these situations in real life. They will also complete a vocabulary task where they will sort word fragments based on type as quickly as they are able. Participants will be asked to return in 24-96 hours for part two where they will repeat a similar scenario reading activity as during time one and fill out a brief questionnaire about your recent behaviors.

ELIGIBILITY:
Inclusion Criteria:

1. Adult aged 18 and older
2. Located in the United States or other primarily English speaking country.
3. Active Amazon Account.

Exclusion Criteria:

* Less than 18 years old.
* Not located in the United States or other primarily English speaking country.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sleep Research Center, Silver Spring, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- HBMT: HBMT: Individual is presented with words with some letters missing and told to complete the word for form non-hostile words.
- Placebo: Alternative to HBMT training. Volunteers is presented with words with some letters missing and told to complete them with whatever comes to mind (no specific instructions).
Period: Overall Study
Arm/Group | HBMT | Placebo
Started | 117 | 112
Completed | 109 | 108
Not Completed | 8 | 4

BASELINE CHARACTERISTICS:
Population: Adults (18 years old or older) in the United States responding to online advertisement on Amazon Mechanical Turk.
Groups:
- Total: Total of all reporting groups
Arm/Group | HBMT | Placebo | Total
Number analyzed (Participants) | 117 | 112 | 229
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Only volunteers who completed all measures were analyzed.
  years
    number analyzed (Participants) | 109 | 108 | 217
    (all) | 40.5 (12.2) | 36.3 (11.4) | 38.4 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Only volunteers who completed all measured wee analyzed/reported. Note: one volunteer refused to report sex.
  Participants
    number analyzed (Participants) | 109 | 107 | 216
    Female | 48 | 49 | 97
    Male | 61 | 58 | 119
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Hostile Attribution Bias
Description: Adapted from the "Angry Cognitions Scale" (Martin and Dahlen 2007). Volunteers read hypothetical scenarios where another person acted aggressively but with unclear intent (e.g., "You are driving through a residential area when someone backs their car out of a driveway and nearly hits you."). Volunteers respond to items (from "Very Unlikely" to "Very Likely") to indicate how they would think about the situation (e.g., "He/she did that just so I'd have to stop. He/she was trying to scare me."). Volunteers responded to one set (4 scenarios) at time point one and a second set (5 scenarios) at time point two. Reponses were summed within each scenario and averaged across scenarios to indicate level of hostile attribution bias. Individual scores at each time point could range from 0 (no hostile attribution bias) to 24 (high hostile attribution bias).
Time Frame: 24-96 hours post HBMT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HBMT | Placebo
Number analyzed (Participants) | 109 | 108
score on a scale | 9.4 (3.9) | 10.8 (3.9)
Statistical Analysis 1: Comparison: HBMT vs Placebo; Test type: Other — Linear Regression; p < .001, Regression, Linear

2. Primary Outcome: Driving Aggression
Description: State Aggression Survey: This survey is adapted from several others in the literature to measure variance along the normal spectrum of aggressive behaviors in daily life that the average person might display (Álvarez-García, et al., 2016; Deffenbacher, et al., 2001; Deffenbacher, J. et al., 2002). The survey specifically asks about driving behaviors (e.g., yelling at other drivers). Scoring is count of aggressive behaviors during reporting period.
Time Frame: 24-96 hours post HBMT
Measure: Mean (Standard Deviation); unit: Number of aggressive driving behaviors
Arm/Group | HBMT | Placebo
Number analyzed (Participants) | 109 | 108
Number of aggressive driving behaviors | 3.0 (3.6) | 3.6 (3.9)
Statistical Analysis 1: Comparison: HBMT vs Placebo; Test type: Other — Regression; p = .027, Regression, Linear

3. Primary Outcome: Aggression On Social Media
Description: Seven items adapted from the Cyber-Aggression Questionnaire for Adolescents by Álvarez-García et al. (2016). Volunteers reported at time point two how often (during preceding 24 h) they engaged in various aggressive online behaviors (e.g., posted rude comments about someone on a social network). Response choices ranged from 1 = never to 4 = always. Scores were recorded dichotomously to represent whether a volunteer reported any online aggression during the reporting period (i.e. "never" was recoded as "0" to indicate no aggression, and all other responses were recoded as "1" to indicate at least some aggression. A higher percentage of volunteers in a study condition reporting usage of aggression on social media indicates a worse outcome for that study condition.
Time Frame: 24-96 hours post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | HBMT | Placebo
Number analyzed (Participants) | 109 | 108
Participants | 15 | 24
Statistical Analysis 1: Comparison: HBMT vs Placebo; Test type: Other — Logistic Regression; p = .004, Regression, Logistic

4. Secondary Outcome: Anger
Description: Trait Anger Scale: Brief measure of trait anger validated by Wilk et al., (2015). Scale (1-5, strongly disagree to strongly agree); Two questions regarding individual's perspective on their anger. Higher values indicate greater anger.
Time Frame: 24-96 hours post HBMT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HBMT | Placebo
Number analyzed (Participants) | 109 | 108
score on a scale | 1.9 (1.1) | 1.7 (.9)

ADVERSE EVENTS:
Time Frame: 24-96 hours
Description: Same definition
Arm/Group | HBMT | Placebo
All-Cause Mortality (participants affected / at risk) | 0/109 | 0/108
Serious Adverse Events (participants affected / at risk) | 0/109 | 0/108
Other Adverse Events (participants affected / at risk) | 0/109 | 0/108

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-16): https://cdn.clinicaltrials.gov/large-docs/40/NCT04015440/Prot_SAP_000.pdf